CLINICAL TRIAL: NCT00187473
Title: Determinants of Disease Severity in Patients With Chronic Hepatitis C and Normal Serum Aminotransferases (Normal Liver Tests)
Brief Title: Natural History of Hepatitis C in Patients With Normal Liver Tests
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: H10102-17633
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Chronic Hepatitis C
Keywords: hepatitis C; HCV; natural history
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: liver biopsy — Liver biopsy every 5 years

SUMMARY:
The Major goals of this project was to assess the natural history of disease in chronic hepatitis C patients with normal ALT and to determine the virologic and host factors associated with disease severity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic hepatitis C and persistently normal liver enzymes
* able to give consent

Exclusion Criteria:

* decompensated liver disease
* any prior antiviral or immunosuppressive therapy
* other liver disease besides hepatitis C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HCV patients with normal ALT
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2000-06 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
ALT | March 2015

CONTACTS AND LOCATIONS:
Overall Officials: Mandana Khalili, MD, Principal Investigator — University of California, San Francisco